CLINICAL TRIAL: NCT06078371
Title: Peri-operative Opioid-free Analgesic Protocol for Orthopedic Trauma Patients
Brief Title: Opioid-Free Pain Treatment in Trauma Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Archie Heddings, MD, Associate Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00149431
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Femoral Neck Fractures; Intertrochanteric Fractures; Femoral Shaft Fracture; Distal Femur Fracture; Patella Fracture; Tibial Shaft Fracture with or Without Associated Fibula Fracture; Ankle Fracture (bimalleolar Equivalent, Bimalleolar, or Trimalleolar); Tibial Pilon Fracture; Talar Head, Neck, Body, or Process Fractures; Calcaneus Fractures; Lisfranc Injuries; Isolated or Multiple Metatarsal Fractures; Phalanx Fractures of the Foot, Single or Multiple; Clavicle Fractures; Proximal Humerus Fractures; Humeral Shaft Fractures; Distal Humerus Fractures (intra or Extra-articular); Olecranon Fractures; Radial Head or Neck Fractures; Elbow Fractures Involving a Combination of Fractures of the Radius and Uln; Forearm Fractures (both Bone Forearm Fractures, Isolated Ulnar Shaft, Isolated Radial Shaft); Distal Radius Fractures
Keywords: Surgical Intervention; Trauma
MeSH Terms: conditions — Femoral Neck Fractures; Hip Fractures; Femoral Fractures, Distal; Patella Fracture; Ankle Fractures; Humeral Fractures, Distal; Olecranon Fracture; Radial Head and Neck Fractures; Wrist Fractures; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The study will be conducted using block randomization, with two six-month blocks of patient enrollment. Block selection will be determined based on the date of the surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid pain treatment (Block 1) (No Intervention): Standard of care pain treatment regimen that involves the use of opioids. Discretion of the medical care team and surgeon will be used for specific opioid pain treatment prescription (quantity, frequency) based on standard of care procedures. All forms of treatment are allowed for the standard of care group which may include but are not limited to blocks, opioids, patient-controlled analgesia, NSAIDs, acetaminophen, muscle relaxing agents, sedation medications, and neuropathic pain medications.
- Opioid-Free pain treatment (Block 2) (Experimental): Pain treatment regiment without the use of opioids. All other pain medication may be used under the discretion of the medical care team and surgeon.
  Interventions: Other: Opioid-free pain treatment

INTERVENTIONS:
Other: Opioid-free pain treatment — Pain treatment includes any medications up to the medical team's discretion aside from opioids.
  Arms: Opioid-Free pain treatment (Block 2)

SUMMARY:
Analgesic drug study that will compare pain outcomes of opioid analgesia and opioid-free analgesia in post-operative orthopedic patients.

DETAILED DESCRIPTION:
This will be a single center randomized trial. The study will be conducted using block randomization, with two six-month blocks of patient enrollment. The first block will consist of patients undergoing treatment of the above-mentioned fractures with normal standard of care pain management protocol (pre-, intra-, and postoperatively). The second block will consist of patients undergoing treatment the same fractures with opioid-free pain management protocol (pre-, intra-, and postoperatively). Block selection will be determined based on the date of the surgery. However, patients initially assigned to the opioid-free protocol that have CKD/laboratory evidence of poor renal function (ie, elevated BUN/Creatinine) or laboratory evidence of liver function issues (ie, cirrhosis, hypoalbuminemia, elevated liver transaminases, elevated GGT) will crossover to the opioid group as NSAID use and acetaminophen use, respectively, are contraindicated. The use of block randomization will preclude the need for the study coordinator to perform any sort of individual randomization or sealed envelope use for treatment assignment. For subjects who meet eligibility criteria, study informed consent will be obtained at the same time as surgical consent. Patients in the standard of care study block will undergo KUMC's normal pain management strategy. Patients in the opioid-free study block will receive the same pain-management drugs as the opioid group aside from receiving opioids; all other medical care will be standard in this group. Postoperative weightbearing, immobilization, perioperative antibiotics, drain usage, and discharge criteria will be determined by institutional protocols and will remain the same for each block. All patients will be started on postoperative chemical anticoagulation prophylaxis as determined by their fracture pattern and medical comorbidities. Patients will be clinically monitored for signs of venous thromboembolism and appropriate diagnostic screening will be utilized as necessary. Wound complications will be monitored by the treating surgeon and managed as necessary. The study team also plans to record patient specific factors including age, sex, BMI, smoking status, comorbidities, and operative time. These variables will be analyzed independently to detect any correlation with the two pain management protocols.

ELIGIBILITY:
Inclusion Criteria:

* Patient is over the age of 18 years old
* Underwent surgical treatment for the injuries of interest (stated elsewhere) by an Orthopedic Traumatology Attending Physician at the University of Kansas Hospital

Exclusion Criteria:

* Patients that are unable to provide informed consent due to sustaining a head injury or incoherence from narcotics given to them post-injury
* Chronic opioid use
* Under the age of 18 years old
* Undergoing revision surgery
* Did not undergo surgical fixation
* Pregnant/nursing women
* Vulnerable populations as defined by the University of Kansas Medical Center IRB
* Did not experience one of the following fractures listed in D.1. above.
* Patients with CKD and/or cirrhosis will be excluded from the opioid-free pain block (block 2) and will only qualify for the standard of care opioid group (Block 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) Pain Scores | From post surgery up until 6 months post surgery
  Patients will be asked how much pain they are experiencing on a 1-10 scale after their surgery. Lower scores mean better outcomes and less pain, higher scores mean worse outcomes.

SECONDARY OUTCOMES:
Postoperative complications | From post surgery up until 6 months post surgery
  Data will be collected on the presence or absence of various complications due to surgery that include: acute kidney injury, subsequent reoperation, amputation, compartment syndrome, surgical site infection, wound dehiscence, nonunion, or venous thromboembolism.
Medication usage (timing) | From post surgery up until 6 months post surgery
  The duration of which analgesia is used to treat post-surgical pain will be measured
Medication usage (quantity) | From post surgery up until 6 months post surgery
  The dosage of analgesia used to treat post-surgical pain will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States